CLINICAL TRIAL: NCT03300960
Title: Usefulness of Medroxyprogesterone Acetate in Follicular Phase in Oocyte Donors.
Brief Title: Usefulness of Medroxyprogesterone Acetate in Follicular Phase in Oocyte Donors. Undergoing Ovarian Stimulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1705-VLC-030-JG
Record Dates: First submitted 2017-09-26; First posted 2017-10-04 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Medroxyprogesterone Acetate; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provera (Experimental)
  Interventions: Drug: Provera 10 mg.
- Orgalutrán Ganirelix (GnRH antagonist) (Active Comparator)
  Interventions: Drug: Ganirelix (GnRH antagonist)

INTERVENTIONS:
Drug: Provera 10 mg. — One 10 mg tablet of MPA (Medroxyprogesterone acetate) is administered every 24 hours from the onset of Controlled Ovarian Stimulation (COS), until the day of triggering.
  Arms: Provera
Drug: Ganirelix (GnRH antagonist) — One ampoule of Ganirelix (GnRH antagonist) a day once diameter of follicles are 14 mm diameter on average until triggering.
  Arms: Orgalutrán Ganirelix (GnRH antagonist)

SUMMARY:
The purpose of this study is to determine whether Medroxyprogesterone Acetate (MPA) administration in follicular phase prevents premature luteinization with equal efficiency as GnRH antagonists and otains similar clinical results in oocyte donation.

DETAILED DESCRIPTION:
Within the new guidelines for stimulation, the use of oral progesterone in follicular phase allows GnRH analogue administration, resulting in greater comfort for patients as well as a reduction in cost. Obtained results are similar to those from conventional protocols in terms of: early luteinization, number of oocytes, embryos number and rate of implantation and gestation or appearance of congenital malformations. Another advantage is the lower incidence of OHSS (Ovarian Hyperstimulation Syndrome).

From a scientific point of view, it would allow a better understanding of folliculogenesis, of progesterone mechanism of action on blocking LH secretion and its effect on ovarian and later embryonic level.

From a clinical point of view, it would simplify COS (Controlled Ovarian Stimulation) by reducing the number of medication administered subcutaneously and their possible side effects on both systemic and local levels. It would be of special interest in 2 groups of patients, for example, oocyte donors and patients undergoing preservation of fertility. To date, there is a lack of studies along these lines.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years (both included)
* Regular Menses (between 25-35 days)
* Absence of physical and psychic pathologies at the time of oocyte donation
* BMI: 18-28 kg(m2 at the time of oocyte donation.
* Other criteria to comply with:

  i. With no relevant personal or family medical history ii. Signing of Informed Consent iii. From a medical point of view:
  1. Healthy ovaries and uterus, with no organic pathology
  2. Ovaries without polycystic aspect
  3. Antral Follicle Count > 12 in the sum of both ovaries
  4. Normal Karyotype
  5. Negative results in infectious illness screening (Hepatitis B Virus; Hepatitis C Virus, VIH Virus Syphilis)
  6. Results within range of general analysis of hemogram, hemostasia y biochemistry.

     Exclusion Criteria:
* Any systemic or metabolic disorder which contraindicate the use of Gonadotrophines
* Medical background of Trombophlebitis or thromboembolic phenomena or Arterial Hypertension
* Severe hepatic insufficiency, cardiovascular illness
* Suspicion or evidence of malignity of mamarian glands or other hormone dependant genital organs
* Known infection of Hepatitis B Virus; Hepatitis C Virus or VIH Virus
* Known hypersensitivity to PMA or its excipients
* Any reason or cause which excluede from the oocyte donation program
* Participation in another clinical trial in the two months prior to the inclusion on this study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 318 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Compare number of oocytes using GnRH antagonist versus PMA. | 36 hours: from triggering until Oocyte retrieval
  Compare oocytes in COS cycles between two groups: using GnRH antagonist versus PMA for avoiding premature luteinization.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Giles, MD PhD, Principal Investigator — Gynecologist IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giles J, Alama P, Gamiz P, Vidal C, Badia P, Pellicer A, Bosch E. Medroxyprogesterone acetate is a useful alternative to a gonadotropin-releasing hormone antagonist in oocyte donation: a randomized, controlled trial. Fertil Steril. 2021 Aug;116(2):404-412. doi: 10.1016/j.fertnstert.2021.02.036. Epub 2021 Apr 2. PMID 33814126